CLINICAL TRIAL: NCT06503770
Title: A Retrospective Chart Review Study of Patients With Chronic Lung Allograft Dysfunction-Bronchiolitis Obliterans Syndrome (CLAD-BOS) Post Lung Transplantation
Status: Completed | Type: Observational
Sponsor: Zambon SpA (Industry)
Responsible Party: Sponsor
Other Study IDs: Z8000N01
Record Dates: First submitted 2024-07-08; First posted 2024-07-16 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Bronchiolitis Obliterans Syndrome Due to and After Lung Transplantation (Disorder)

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The aim of this study is to describe the forced expiratory volume in 1 second (FEV1) decline and natural disease evolution in patients affected by CLAD-BOS after lung transplantation and receiving an immunosuppressive therapy as standard of care.

DETAILED DESCRIPTION:
This is a retrospective, multinational, multicenter chart review study of adult patients with clinically diagnosed CLAD-BOS after lung transplantation. All data will be retrospectively collected from patient records starting from lung transplantation date through last date of available data, and as such, no interventions will be applied as part of this study.

The observational period for each patient will be from lung transplant date until last date of data available or death, whichever occurs earlier and will include the following time periods:

Diagnosis window: 01 January 2013 through most recent data available.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients ≥ 18 years of age on the date of CLAD-BOS diagnosis
2. Patients with a CLAD-BOS clinician diagnosis from as early as 01 January 2013
3. Patients with CLAD-BOS clinician diagnosis made at least 12 months after lung transplant
4. Patients received at least basic maintenance regimen of immunosuppressive agents including tacrolimus, a second agent such as but not limited to mycophenolate mofetil or azathioprine (or other anti-proliferative agent), and a systemic corticosteroid such as prednisone as third agent for at least 1 month before the index date. As long as the basic maintenance regimen is maintained for the abovementioned period, patients will still be considered eligible for the study even if they are receiving other immunosuppressive agents in addition to the basic maintenance regimen.

Exclusion Criteria:

1. Patients with severe concomitant disease at the time of index date, which according to physician's judgment, can interfere with CLAD-BOS progression and mortality (e.g., malignancies, severe chronic diseases)
2. Patients who have been exposed to any investigational medical products in the 4 weeks prior to index date or during the post-diagnosis period
3. Patients with confirmed other CLAD phenotype (e.g., restrictive allograft syndrome) according to physician's judgment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will include adult patients aged ≥ 18 years who are recipients of a lung transplant and diagnosed with CLAD-BOS from the first of January 2013 following transplantation.
Sampling Method: Probability Sample
Enrollment: 284 (Actual)
Dates: Start 2024-06-27 (Actual); Primary Completion 2025-04-02 (Actual); Study Completion 2025-04-02 (Actual)

PRIMARY OUTCOMES:
To evaluate the FEV1 trajectory of patients diagnosed with CLAD-BOS | Up to 12 years
  Change in FEV1 trajectory over time

CONTACTS AND LOCATIONS:
Overall Officials: Bucchioni, MD, Study Director — Zambon SpA
Locations (6):
- United States (3):
  - Cleveland Clinic Main Campus, Cleveland, Ohio
  - Baylor Scott and White Health Advanced Lung Disease Specialists, Columbus, Ohio
  - Baylor Scott and White Health Advanced Lung Disease Specialists, Dallas, Texas
- Universitaire Ziekenhuizen Leuven (UZ Leuven) Campus Gasthuisberg, Leuven, Leuven, Belgium
- Spain (2):
  - Hospital Universitario Reina Sofia, Córdoba, Andalusia
  - Universidad de Cantabria (UC) Hospital Universitario Marques de Valdecilla (HUMV), Santander, Cantabria

IPD SHARING:
Plan to Share IPD: No